CLINICAL TRIAL: NCT04988087
Title: A Multi-center, Randomized, Participant- and Investigator- Blinded, Placebo-controlled, Parallel Group Basket Study to Evaluate the Safety, Tolerability and Efficacy of MHV370 in Participants With Sjögren's Syndrome or Mixed Connective Tissue Disease
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of MHV370 in Participants With Sjogren's Syndrome (SjS) or Mixed Connective Tissue Disease (MCTD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMHV370A12201; 2020-004937-19 (EudraCT Number)
Record Dates: First submitted 2021-07-26; First posted 2021-08-03 (Actual); Results first posted 2024-07-08 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Sjogren Syndrome; Mixed Connective Tissue Disease
Keywords: Sicca Syndrome; Sjogren Syndrome; Connective Tissue Disease, Mixed; MCTD; Sharp Syndrome
MeSH Terms: conditions — Sjogren's Syndrome; Mixed Connective Tissue Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SjS participants: MHV370 (Experimental): SjS participants randomized in the MHV370 arm will be treated with MHV370 for 24 weeks. Double-blind supply will be used.
  Interventions: Drug: MHV370
- SjS participants: Placebo (Placebo Comparator): SjS participants randomized in the placebo arm will be treated with placebo for 24 weeks. Double-blind supply will be used.
  Interventions: Drug: Placebo
- MCTD participants: MHV370 (Experimental): MCTD participants randomized in the MHV370 arm will be treated with MHV370 for 24 weeks. Double-blind supply will be used.
  Interventions: Drug: MHV370
- MCTD participants: Placebo (Placebo Comparator): MCTD participants randomized in the placebo arm will be treated with placebo for 24 weeks. Double-blind supply will be used.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MHV370 — MHV370 for 24 weeks
  Arms: MCTD participants: MHV370; SjS participants: MHV370
Drug: Placebo — Placebo for 24 weeks
  Arms: MCTD participants: Placebo; SjS participants: Placebo

SUMMARY:
This study was a basket trial designed to establish safety, tolerability and efficacy of MHV370 in Sjögren's Syndrome (SjS) and Mixed Connective Tissue Disease (MCTD).

DETAILED DESCRIPTION:
This was a randomized, participant and investigator blinded, placebo-controlled, multi center parallel group basket study to evaluate the safety, tolerability and efficacy of MHV370 in participants with Sjögren's Syndrome (SjS) or with Mixed Connective Tissue Disease (MCTD). Participants first underwent a screening period of up to 6 weeks, followed by a treatment duration of 24 weeks and a follow-up period of 4 weeks. Total study duration for each participant was up to 34 weeks. Participants with SjS were randomized in a 1:1 ratio to MHV370 or placebo and participants with MCTD were randomized in a 1:1 ratio to MHV370 or placebo.

ELIGIBILITY:
Inclusion Criteria:

SjS and MCTD:

• Fully vaccinated with any locally approved COVID-19 vaccination including booster vaccinations if required by local guidelines

SjS:

* Unstimulated whole salivary flow rate of > 0 mL/min at screening
* Classification of Sjögren's Syndrome according to the 2016 ACR/EULAR criteria at screening
* Screening ESSDAI (based on weighted score) ≥ 5 from 8 defined domains (biologic, hematologic, articular, cutaneous, glandular, lymphadenopathy, renal, constitutional).

MCTD:

* Diagnosis of MCTD based on criteria like a) Raynaud's phenomenon b) At least two of the four following signs: i) synovitis, ii) myositis, iii) swollen fingers and vi) interstitial lung disease
* Patients with overlap syndromes, i.e. patients meeting diagnostic criteria for systemic autoimmune disease other than MCTD may be included unless they have major organ involvement as judged by the investigator

Exclusion Criteria:

SjS and MCTD:

* Prior use of B-cell depleting therapy within 6 months of baseline. For participants who received B-cell depleting therapy within 6 -12 months of baseline visit, B-cell count should be within normal range
* Prior treatment with any of the following within 3 months of baseline: CTLA4-Fc Ig (abatacept), Anti-TNF mAb, Intravenous Ig, Plasmapheresis, i.v. or oral cyclophosphamide, i.v. or oral cyclosporine A
* Screening CBC laboratory values as follows: Hemoglobin levels < 8 g/dL (< 5 mmol/L), Total leukocyte count < 2,000/µL (2 x 109/L), Platelets < 50,000/µL (50 x 109/L), Neutrophil count < 1,000/µL (1 x 109/L)
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they use a highly effective method of contraception

SjS:

* Sjögren's Syndrome overlap syndromes where another autoimmune disease constitutes the primary illness
* Required regular use of medications known to cause, as a major side effect, dry mouth / eyes

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- China (2):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Changchun, Jilin
- Novartis Investigative Site, Berlin, Germany
- Hungary (2):
  - Novartis Investigative Site, Székesfehérvár, Fejér
  - Novartis Investigative Site, Debrecen
- Poland (3):
  - Novartis Investigative Site, Bialystok, Podlaskie Voivodeship
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
- Novartis Investigative Site, Madrid, Spain
- Novartis Investigative Site, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Raaphorst J, Gullick NJ, Shokraneh F, Brassington R, Min M, Ali SS, Gordon PA. Non-targeted immunosuppressive and immunomodulatory therapies for idiopathic inflammatory myopathies. Cochrane Database Syst Rev. 2025 Aug 11;8(8):CD015855. doi: 10.1002/14651858.CD015855. PMID 40787733
- [Derived] Raaphorst J, Gullick NJ, Shokraneh F, Brassington R, Min M, Ali SS, Gordon PA. Targeted immunosuppressive and immunomodulatory therapies for idiopathic inflammatory myopathies. Cochrane Database Syst Rev. 2025 Aug 1;8(8):CD015854. doi: 10.1002/14651858.CD015854. PMID 40747756
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1877

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 10 investigative sites in 6 countries/regions.
Pre-assignment Details: There was a screening period of up to 6 weeks to assess participants eligibility.
Groups:
- MHV370 200mg - SjS: MHV370 200mg oral dose, twice daily. SjS participants.
- Placebo - SjS: Placebo oral dose, twice daily. SjS participants.
- MHV370 200mg - MCTD: MHV370 200mg oral dose, twice daily. MCTD participants.
- Placebo - MCTD: Placebo oral dose, twice daily. MCTD participants.
Period: Overall Study
Arm/Group | MHV370 200mg - SjS | Placebo - SjS | MHV370 200mg - MCTD | Placebo - MCTD
Started | 12 | 14 | 2 | 2
Completed | 0 | 4 | 1 | 0
Not Completed | 12 | 10 | 1 | 2
Not completed — Adverse Event | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Technical problems | 7 | 9 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MHV370 200mg - SjS | Placebo - SjS | MHV370 200mg - MCTD | Placebo - MCTD | Total
Number analyzed (Participants) | 12 | 14 | 2 | 2 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (12.20) | 54.7 (9.67) | 35.0 (12.73) | 44.0 (0.00) | 50.5 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 2 | 2 | 30
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 3 | 0 | 0 | 6
  White | 9 | 11 | 2 | 2 | 24

OUTCOME MEASURES:

1. Primary Outcome: SjS Participants: Change From Baseline in Eular Sjögren's Disease Activity Index (ESSDAI) After 24 Weeks of Treatment
Description: The ESSDAI is an established disease outcome measure for Sjögren's syndrome that classifies disease activity in 3-4 levels according to their severity (i.e., no, low, moderate, high), over each of 12 organ-specific domains. These scores are then summed across the 12 domains in a weighted manner to provide the total score. The score range is 0 - 123, where a higher ESSDAI score indicates more severe symptoms. A negative change score from baseline indicates improvement.
Time Frame: Baseline, Week 24
Population: The pharmacodynamic (PD) analysis set included all participants who received any study drug and had no protocol deviations with relevant impact on PD/efficacy data. The data includes only participants who completed Week 24. Only participants with evaluable records are included.
Measure: Mean (Standard Error); unit: Score on scale
Arm/Group | MHV370 200mg - SjS | Placebo - SjS
Number analyzed (Participants) | 0 | 4
Score on scale |  | -4.39 (2.41)

2. Primary Outcome: MCTD Participants: Change From Baseline in Physician's Global Assessment Scale (PhGA) After 24 Weeks of Treatment
Description: The physician's global assessment scale is used for the Investigator to rate the disease activity of their patient using 100 mm visual analog scale (VAS) ranging from "no disease activity" (0) to "maximal disease activity" (100). A negative change score from baseline indicates improvement. Only participants with evaluable records are included.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Median (Full Range); unit: Score on scale
Arm/Group | MHV370 200mg - MCTD | Placebo - MCTD
Number analyzed (Participants) | 1 | 0
Score on scale | -62.00 [-62.00 to -62.00] |

3. Secondary Outcome: SjS and MCTD Participants: Maximum Observed Plasma Concentrations (Cmax) of MHV370 at Steady State
Description: Cmax is the maximum (peak) observed plasma concentration of MHV370 after single dose administration. Pharmacokinetic (PK) parameters were calculated based on MHV370 plasma concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC-MS/MS) method with a lower limit of quantification of 1.0 ng/mL. Cmax was determined using non-compartmental methods.
Time Frame: pre-dose, 0.5, 1, 2 ,4 and 6 hours after dosing at week 4
Population: The pharmacokinetic (PK) analysis set included participants with at least one available valid (i.e., not flagged for exclusion) PK concentration measurement, who received MHV370 and with no protocol deviations with impact on PK data. Only participants with evaluable records are included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MHV370 200mg - SjS | MHV370 200mg - MCTD
Number analyzed (Participants) | 8 | 1
ng/mL | 278 (85.7) | 194

4. Secondary Outcome: SjS and MCTD Participants: Area Under the Plasma Concentration-time Curve From Time Zero to 6 Hours (AUC0-6h) of MHV370
Description: The AUC from time zero to the 6-hours post-dose sampling time. Pharmacokinetic (PK) parameters were calculated based on MHV370 plasma concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC-MS/MS) method with a lower limit of quantification of 1.0 ng/mL. AUClast was determined using non-compartmental methods.
Time Frame: pre-dose, 0.5, 1, 2 ,4 and 6 hours after dosing at week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | MHV370 200mg - SjS | MHV370 200mg - MCTD
Number analyzed (Participants) | 5 | 1
ng*h/mL | 1060 (462) | 742

5. Secondary Outcome: SjS and MCTD Participants: Time to Reach Maximum Plasma Concentrations (Tmax) of MHV370 at Steady State
Description: Tmax is the time to reach maximum (peak) plasma concentration of MHV370 after single dose administration. Pharmacokinetic (PK) parameters were calculated based on MHV370 plasma concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC-MS/MS) method with a lower limit of quantification of 1.0 ng/mL. Tmax was determined using non-compartmental methods.
Time Frame: pre-dose, 0.5, 1, 2 ,4 and 6 hours after dosing at week 4
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Groups:
- MHV370 200mg - MCTD: MHV370 200mg oral dose, twice daily. - MCTD participants
Arm/Group | MHV370 200mg - SjS | MHV370 200mg - MCTD
Number analyzed (Participants) | 8 | 1
hours | 1.50 [1.00 to 4.00] | 2.00

6. Secondary Outcome: SjS and MCTD Participants: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale
Description: The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F v4) is a short, 13-item patient-reported measure, easy-to-administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a 5-point Likert scale (0 = not at all, 1 = a little bit, 2 = somewhat, 3 = quite a bit, 4 = very much). To score the FACIT-fatigue, all items are summed to create a single fatigue score with a range from 0 to 52, where a higher FACIT-F score indicates more severe symptoms. A negative change score from baseline indicates improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 20 and 24
Population: The pharmacodynamic (PD) analysis set included all participants who received any study drug and had no protocol deviations with relevant impact on PD/efficacy data. Data from participants who have discontinued treatment early are regarded as missing after the treatment discontinuation. Only participants with evaluable records are included.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | MHV370 200mg - SjS | Placebo - SjS | MHV370 200mg - MCTD | Placebo - MCTD
Number analyzed (Participants) | 8 | 12 | 2 | 1
Score on scale
  Week 4 | 0.13 (3.271) | -1.58 (6.052) | 15.50 (9.192) | -3.00
  Week 8: number analyzed (Participants) | 7 | 10 | 2 | 1
  Week 8 | 3.14 (5.928) | -2.80 (4.185) | 20.00 (7.071) | -2.00
  Week 12: number analyzed (Participants) | 4 | 7 | 1 | 0
  Week 12 | -1.25 (6.702) | 2.71 (8.826) | 20.00 |
  Week 20: number analyzed (Participants) | 1 | 5 | 1 | 0
  Week 20 | -9.42 | 4.80 (8.758) | 23.00 |
  Week 24: number analyzed (Participants) | 0 | 4 | 1 | 0
  Week 24 |  | 5.75 (10.782) | 30.00 |

7. Secondary Outcome: SjS and MCTD Participants: Change From Baseline in Physician Global Assessment (PhGA)
Description: The physician's global assessment scale is used for the Investigator to rate the disease activity of their patient using 100 mm visual analog scale (VAS) ranging from "no disease activity" (0) to "maximal disease activity" (100). A negative change score from baseline indicates improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 20 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | MHV370 200mg - SjS | Placebo - SjS | MHV370 200mg - MCTD | Placebo - MCTD
Number analyzed (Participants) | 8 | 12 | 2 | 1
Score on scale
  Week 4 | -1.75 (12.658) | -5.25 (11.185) | -20.50 (12.021) | -15.00
  Week 8: number analyzed (Participants) | 7 | 10 | 2 | 1
  Week 8 | 2.57 (12.608) | -8.90 (11.474) | -39.00 (18.385) | -12.50
  Week 12: number analyzed (Participants) | 4 | 7 | 1 | 0
  Week 12 | -4.00 (20.559) | -19.43 (14.328) | -66.00 |
  Week 20: number analyzed (Participants) | 1 | 5 | 1 | 0
  Week 20 | 3.00 | -14.60 (22.423) | -64.00 |
  Week 24: number analyzed (Participants) | 0 | 4 | 1 | 0
  Week 24 |  | -30.75 (19.534) | -62.00 |

8. Secondary Outcome: SjS Participants: Change From Baseline in Eular Sjögren's Syndrome Disease Activity Index (ESSDAI)
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 20 and 24
Population: The pharmacodynamic (PD) analysis set included all participants who received any study drug and had no protocol deviations with relevant impact on PD/efficacy data. Only participants with evaluable records are included.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | MHV370 200mg - SjS | Placebo - SjS
Number analyzed (Participants) | 8 | 12
Score on scale
  Week 4 | -0.25 (1.753) | -3.67 (9.355)
  Week 8: number analyzed (Participants) | 7 | 10
  Week 8 | 0.57 (6.528) | -4.80 (11.487)
  Week 12: number analyzed (Participants) | 3 | 7
  Week 12 | -3.00 (4.583) | -3.43 (7.656)
  Week 20: number analyzed (Participants) | 1 | 5
  Week 20 | -2.00 | 0.00 (14.629)
  Week 24: number analyzed (Participants) | 0 | 4
  Week 24 |  | -0.25 (11.117)

9. Secondary Outcome: SjS Participants: Change From Baseline in Eular Sjögren's Syndrome Patient Reported Index (ESSPRI)
Description: The ESSPRI is an established disease outcome measure for Sjögren's syndrome. The ESSPRI is a patient-reported, subjective symptom index which consists of three questions covering the cardinal symptoms of Sjögren's syndrome: dryness, fatigue and pain (articular and/or muscular). The participant can assess severity of symptoms they experience on a single numerical scale of 0-10 (0 =no symptom at all and 10 = worst symptom imaginable) for each of the three domains. The overall ESSPRI score is calculated as the mean of the three individual domains where all domains carry the same weight. Minimum score can be 0 and maximum score can be 10, where a higher ESSPRI score indicates more severe symptoms. A negative change score from baseline indicates improvement.
Time Frame: baseline, weeks 4, 8, 12, 20 and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | MHV370 200mg - SjS | Placebo - SjS
Number analyzed (Participants) | 8 | 12
Score on scale
  Week 4 | -0.12 (0.354) | -0.53 (1.105)
  Week 8: number analyzed (Participants) | 7 | 10
  Week 8 | -0.67 (0.793) | -0.37 (1.511)
  Week 12: number analyzed (Participants) | 4 | 7
  Week 12 | -0.42 (0.500) | -1.38 (1.976)
  Week 20: number analyzed (Participants) | 1 | 5
  Week 20 | -0.17 | -2.20 (1.865)
  Week 24: number analyzed (Participants) | 0 | 4
  Week 24 |  | -2.00 (2.000)

10. Secondary Outcome: SjS Participants: Change From Baseline to the Salivary Flow Rate
Description: Unstimulated whole salivary fluid secretions were collected over 5 minutes from participants. All assessments were performed at a fixed time of the day to minimize fluctuations related to the circadian rhythm of salivary flow and composition. Participants were instructed not to eat, drink or smoke for 90 minutes before the assessment. The start time and end time of saliva collection were recorded to calculate the salivary flow rate per minute. Only participants with evaluable records are included.
Time Frame: Baseline, Weeks 4, 12 and 24
Population: The pharmacodynamic (PD) analysis set included all participants who received any study drug and had no protocol deviations with relevant impact on PD/efficacy data.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | MHV370 200mg - SjS | Placebo - SjS
Number analyzed (Participants) | 12 | 14
mL/min
  Week 4: number analyzed (Participants) | 8 | 12
  Week 4 | 0.162 (0.2735) | -0.127 (0.7914)
  Week 12: number analyzed (Participants) | 4 | 7
  Week 12 | 0.144 (0.2109) | 0.183 (0.3944)
  Week 24: number analyzed (Participants) | 0 | 4
  Week 24 |  | 0.564 (0.9193)

11. Secondary Outcome: SjS Participants: Change From Baseline to the Schirmer's Test
Description: Schirmer's test is used to determine whether the eye produces enough tears to keep it moist especially for those who suffer from dry eye syndrome. A strip is placed in the lower eyelid for 5 minutes to assess tear production. After 5 minutes, the filter paper is removed and the distance between the leading edge of wetness and the initial fold is measured, using a millimeter ruler. Tear deficiency is defined as <5 mm wetting of the paper after 5 minutes.
Time Frame: Baseline, Week 4, 12 and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milimeter
Arm/Group | MHV370 200mg - SjS | Placebo - SjS
Number analyzed (Participants) | 12 | 14
milimeter
  Week 4, right eye: number analyzed (Participants) | 8 | 12
  Week 4, right eye | -1.5 (4.87) | 0.0 (3.59)
  Week 12, right eye: number analyzed (Participants) | 4 | 7
  Week 12, right eye | -1.0 (2.16) | 5.3 (8.81)
  Week 24, right eye: number analyzed (Participants) | 0 | 4
  Week 24, right eye |  | -3.0 (6.32)
  Week 4, left eye: number analyzed (Participants) | 8 | 12
  Week 4, left eye | 1.1 (1.96) | 1.6 (6.01)
  Week 12, left eye: number analyzed (Participants) | 4 | 7
  Week 12, left eye | 2.0 (1.83) | 4.9 (12.50)
  Week 24, left eye: number analyzed (Participants) | 0 | 4
  Week 24, left eye |  | -1.0 (2.94)

12. Secondary Outcome: SjS Participants: Sjögren's Tool for Assessing Response (STAR) Response Over Time up to Week 24
Description: STAR is a composite responder index, including in a single tool all main disease features, and designed for use as a key efficacy endpoint in SjS Domain Point Definition of response.
  Points are assigned in the following 5 domains, if the corresponding criteria are met:
  * Systemic activity, if decrease in clin ESSDAI ≥ 3 points: 3 points
  * Patient reported outcome, if decrease in ESSPRI ≥ 1 point or 15%: 3 points
  * Lacrimal gland function (assessed by Schirmer's test), if abnormal score at baseline: increase ≥ 5 mm from baseline OR if normal score at baseline: no change to abnormal: 1 point
  * Salivary gland function (assessed by unstimulated salivary flow), if increase ≥ 25% from baseline: 1 point
  * Biological (assessed by serum IgG levels), if decrease ≥ 10%: 1 point The Total Score is the sum of all 5 domain scores, ranging from 0 to 9 points. A STAR responder is defined as ≥ 5 points in the Total Score.
Time Frame: Baseline, Week 4, 12 and 24
Population: The pharmacodynamic (PD) analysis set included all participants who received any study drug and had no protocol deviations with relevant impact on PD/efficacy data. Missing responses will be treated as non-responders. Only participants with evaluable records are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MHV370 200mg - SjS | Placebo - SjS
Number analyzed (Participants) | 12 | 14
Participants
  Week 4 | 0 | 3
  Week 12 | 1 | 4
  Week 24 | 0 | 2

13. Secondary Outcome: MCTD: Change From Baseline in Articular and Pulmonary Domains of the Eular Sjögren's Syndrome Disease Activity Index (ESSDAI)
Description: The ESSDAI is an established disease outcome measure for Sjögren's syndrome that classifies disease activity in 3-4 levels according to their severity (i.e., no, low, moderate, high), over each of 12 organ-specific domains. Participants with Mixed Connective Tissue Disease (MCTD) completed the articular (from 0 "no activity" to 3 "high activity") and pulmonary (from 0 "no activity to 3 "high activity") domains of the ESSDAI only. For MCTD participants, the score range is 0-21, where a higher score indicates more severe symptoms. A negative change score from baseline indicates improvement.
Time Frame: Baseline, Weeks 4, 8, 12 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | MHV370 200mg - MCTD | Placebo - MCTD
Number analyzed (Participants) | 2 | 1
Score on scale
  Week 4 - articular | 0.00 (0.000) | 0.00
  Week 8 - articular | -1.00 (0.000) | 0.00
  Week 12 - articular: number analyzed (Participants) | 1 | 0
  Week 12 - articular | -1.00 |
  Week 24 - articular: number analyzed (Participants) | 1 | 0
  Week 24 - articular | -2.00 |
  Week 4 - pulmonary | 0.00 (0.000) | 0.00
  Week 8 - pulmonary | -0.50 (0.707) | 0.00
  Week 12 - pulmonary: number analyzed (Participants) | 1 | 0
  Week 12 - pulmonary | -1.00 |
  Week 24 - pulmonary: number analyzed (Participants) | 1 | 0
  Week 24 - pulmonary | -1.00 |

14. Secondary Outcome: MCTD Participants: Change From Baseline in Forced Vital Capacity (FVC)
Description: Forced Vital Capacity (FVC) is the total amount of air exhaled during the Forced expiratory volume (FEV) test measured through spirometry testing. FEV measures how much air a person can exhale during a forced breath. A positive change from baseline is considered a favorable outcome.
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: liters (L)
Arm/Group | MHV370 200mg - MCTD | Placebo - MCTD
Number analyzed (Participants) | 1 | 0
liters (L) | 0.530 |

15. Secondary Outcome: MCTD Participants: Change From Baseline in Forced Expiratory Volume During the First Second (FEV1) of a Forced Breath
Description: FEV1 (forced expiratory volume in one second) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing. A positive change from baseline in FEV1 is considered a favourable outcome.
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: liters (L)
Arm/Group | MHV370 200mg - MCTD | Placebo - MCTD
Number analyzed (Participants) | 1 | 0
liters (L) | 0.250 |

16. Secondary Outcome: MCTD Participants: Change From Baseline in Forced Expiratory Volume During the First Two Seconds (FEV2) of a Forced Breath
Description: FEV2 (forced expiratory volume in two seconds) is the amount of air which can be forcibly exhaled from the lungs in the first two seconds of a forced exhalation, measured through spirometry testing. A positive change from baseline in FEV2 is considered a favourable outcome.
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: liters (L)
Arm/Group | MHV370 200mg - MCTD | Placebo - MCTD
Number analyzed (Participants) | 1 | 0
liters (L) | 0.410 |

17. Secondary Outcome: MCTD Participants: Change From Baseline in Forced Expiratory Volume During the First Three Seconds (FEV3) of a Forced Breath
Description: FEV3 (forced expiratory volume in three seconds) is the amount of air which can be forcibly exhaled from the lungs in the first three seconds of a forced exhalation, measured through spirometry testing. A positive change from baseline in FEV3 is considered a favourable outcome.
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: liters (L)
Arm/Group | MHV370 200mg - MCTD | Placebo - MCTD
Number analyzed (Participants) | 1 | 0
liters (L) | 0.460 |

18. Secondary Outcome: MCTD Participants: Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO)
Description: Diffusing capacity of the lungs for carbon monoxide (DLCO) is a measurement to assess the ability of the lungs to transfer gas from inspired air to the bloodstream. Inhaled carbon monoxide (CO) is used for this test due to its high affinity for hemoglobin. During a ten-second breath-hold, DLCO measures uptake of CO per time per CO pressure. The outcome is presented as percentage of predicted DLCO value.
Time Frame: Baseline, Week 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of predicted DLCO
Arm/Group | MHV370 200mg - MCTD | Placebo - MCTD
Number analyzed (Participants) | 1 | 2
percentage of predicted DLCO
  Baseline | 84.0 | 95.5 (2.12)
  Week 24: number analyzed (Participants) | 0 | 0

19. Secondary Outcome: MCTD Participants: Change From Baseline in King's Brief Interstitial Lung Disease (K-BILD)
Description: The K-BILD questionnaire is a self-administered health-status questionnaire that has been developed in patients with interstitial lung diseases. It consists of 15 items in three domains: breathlessness and activities, psychological factors, and chest symptoms. Total scores range from 0 to 100, with higher scores representing better health status.
Time Frame: Baseline, Weeks 4, 8, 12 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | MHV370 200mg - MCTD | Placebo - MCTD
Number analyzed (Participants) | 2 | 1
Score on scale
  Week 4 | 3.00 (4.243) | -2.00
  Week 8 | 13.00 (9.899) | 0.00
  Week 12: number analyzed (Participants) | 1 | 0
  Week 12 | 21.00 |
  Week 24: number analyzed (Participants) | 1 | 0
  Week 24 | 58.00 |

20. Secondary Outcome: MCTD Participants: Change From Baseline in Raynaud's Condition Score (RCS)
Description: The Raynaud's Condition score (RCS) is participant's rating of difficulty considering number of attacks, duration, amount of pain, numbness, or other symptoms caused in the fingers (including painful sores) due to the Raynaud's phenomenon and impact of Raynaud's alone on use of hands every day. An 11-point Likert scale is used to rate the difficulty caused by the condition with 0 = no difficulty and 10 = extreme difficulty. Participants are asked to select the number that best describes their difficulty, with higher score indicating worse condition.
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | MHV370 200mg - MCTD | Placebo - MCTD
Number analyzed (Participants) | 2 | 2
Score on scale
  Week 4: number analyzed (Participants) | 2 | 1
  Week 4 | -2.50 (3.536) | 1.00
  Week 12: number analyzed (Participants) | 1 | 0
  Week 12 | -1.00 |
  Week 24: number analyzed (Participants) | 1 | 0
  Week 24 | -2.00 |

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of approximately 199 days.
Groups:
- sjs_MHV: sjs_MHV
- sjs_Placebo: sjs_Placebo
- MCTD_MHV: MCTD_MHV
- MCTD_Placebo: MCTD_Placebo
- Total: Total
Arm/Group | sjs_MHV | sjs_Placebo | MCTD_MHV | MCTD_Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14 | 0/2 | 0/2 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14 | 0/2 | 1/2 | 1/30
Other Adverse Events (participants affected / at risk) | 12/12 | 12/14 | 1/2 | 2/2 | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | sjs_MHV (N=12) | sjs_Placebo (N=14) | MCTD_MHV (N=2) | MCTD_Placebo (N=2) | Total (N=30)
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | sjs_MHV (N=12) | sjs_Placebo (N=14) | MCTD_MHV (N=2) | MCTD_Placebo (N=2) | Total (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 3
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 3
Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1
Thyroid mass (Endocrine disorders) | 1 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 1
Conjunctival suffusion (Eye disorders) | 1 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 2
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Mouth swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1
Swelling (General disorders) | 1 | 0 | 0 | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 1 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 4 | 2 | 0 | 0 | 6
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Dacryocanaliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 1 | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Antinuclear antibody increased (Investigations) | 0 | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 1
Complement factor C3 decreased (Investigations) | 0 | 2 | 0 | 0 | 2
Complement factor C4 decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 2
Facial paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 4 | 0 | 2 | 8
Hypergeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT04988087/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT04988087/SAP_001.pdf